CLINICAL TRIAL: NCT03579550
Title: The Comparison of Reproductive Outcomes of Hsyteroscopic Metroplasty Versus Spontaneous Coitus Plus COH/IUI Cycles in Unexplained Infertile Women With Dysmorphic Uterus
Brief Title: Hysteroscopic Metroplasty in Unexplained Infertile Women With Dysmorphic Uterus
Acronym: COH/IUI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bulent Haydardedeoglu (Other)
Responsible Party: Sponsor-Investigator, Bulent Haydardedeoglu, Associate Prof. M.D., Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA17/151
Record Dates: First submitted 2018-06-26; First posted 2018-07-06 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Hysteroscopy; Pregnancy Rate; Abortion; Ectopic Pregnancy; Intrauterine Insemination
Keywords: dysmorphic uterus, metroplasty, hysteroscopy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Intervention Model Description: prospective randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm: Hysterocopy group (Active Comparator): Office hyteroscopic metroplasty will be performed. After oparetion 9 months spontaneous conception Intervention arm for hysteroscopy group
  Interventions: Procedure: office hysteroscopic metroplasty intervention arm
- Spontaneous cycles plus COH/IUI (No Intervention): Six months spontaneous coitus cycles plus 3 cycles of Clomiphene citrate and intrauterine insemination (COH/IUI)

INTERVENTIONS:
Procedure: office hysteroscopic metroplasty intervention arm — One group will be performed hysteroscopic metroplasty Second group will be undertaken to six months spontaneous coitus and three cycles of COH/IUI
  Other Names: spontaneous coitus plus COH/IUI
  Arms: Intervention arm: Hysterocopy group

SUMMARY:
The correlation between dysmorphic uterus and infertility still remains enigmatic. We aim to evaluate the reproductive outcomes of metroplasty via office hysteroscopy in unexplained infertile women with dysmorphic uterus with comparing a group of unexplained infertile women performing 6 months spontaneous cycles plus 3 cycles controlled ovarian hyperstimulation and intrauterine insemination by randomized trial.

DETAILED DESCRIPTION:
A dysmorphic uterus is a second-class (Class U1) uterine anomaly in the The European Society of Human Reproduction and Embryology (ESHRE) and the European Society for Gynaecological Endoscopy (ESGE) (ESHRE/ESGE) consensus on the classification of congenital genital tract anomalies, which was formerly known as "T-shaped uterus" in the American Fertility Society (AFS) Classification of Anomalies of the Müllerian Duct that leads to poor reproductive and obstetric outcomes.

The reproductive performance of dysmorphic uterus is not well-known issue. We designed a randomized trial in unexplained infertile couples women with dysmorphic uterus. After allocation of properly selected women, hysteroscopy group will be undertaken metroplasty procedure and 9 months follow-up period with natural conception. Second group will be undertaken to six months spontaneous coitus and three cycles clomiphene citrate and intrauterine insemination cycles. After nine months of follow-up of both groups, the pregnancy and reproductive outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Unexplained infertile couples with;

1. Dysmorpic uterus in hysterosalpingography
2. Normal spermiogram

2. Bilateral patent tubes in hysterosalpingography 3. Normal ovarian reserve (AMH >1.5 ng/dl and/or total bilateral antral follicle count >8)

Exclusion Criteria:

1. Women with history of pelvic surgery including endometriosis and/or tubal surgery
2. women with endometrioma which was visualised/suspected on transvaginal ultrasonography
3. Women with anovulation
4. Women with diminished ovarian reserve (AMH < 1.5 ng/dl and/or total bilateral antral follicle count <8)
5. Couples with abnormal spermiogram parameters (oligospermia, oligoasthenospermia, oligoasthenoteratozoospermia, azospermia)
6. Women with alive children
7. Obese women (BMI>30 kg/m2)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with dysmorphic uterus
Enrollment: 86 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate (CPR) | 9 months
  Intrauterine gestational sac with viable fetal heart rate

SECONDARY OUTCOMES:
abortion | 10 weeks
  the loss of pregnancy
ectopic pregnancy rate | 10 weeks
  gestation with out of uterine cavity

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Haydardedeoglu, Assoc.Prof., Principal Investigator — Baskent University
Locations (1):
- Bulent Haydardedeoglu, Adana, Turkey (Türkiye)